CLINICAL TRIAL: NCT04243395
Title: Effects of Consuming Ounce Equivalent Portions of Fresh Pork Versus Nuts, Beans, and Eggs, as Defined by the Dietary Guidelines for Americans on Essential Amino Acid Substrate Availability for Protein Anabolism in Older Adults
Brief Title: Protein Source on Plasma Amino Acid Concentrations In Older Adults
Acronym: S55
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Principal Investigator, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: IRB-2019-354
Record Dates: First submitted 2020-01-18; First posted 2020-01-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Protein Deposition
MeSH Terms: interventions — Pork Meat; Eggs

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pork (Experimental): 1 ounce lean pork
  Interventions: Other: Pork
- Egg (Experimental): 1 large whole egg
  Interventions: Other: Egg
- Black beans (Experimental): 0.5 cups of cooked black beans
  Interventions: Other: Black beans
- Almonds (Experimental): 0.5 ounce of whole almonds
  Interventions: Other: Almonds

INTERVENTIONS:
Other: Pork — 1 oz lean pork
  Arms: Pork
Other: Egg — 1 large whole egg
  Arms: Egg
Other: Black beans — 0.5 cups cooked black beans
  Arms: Black beans
Other: Almonds — 0.5 oz almonds
  Arms: Almonds

SUMMARY:
This study will determine the effect of the same ounce-equivalents of fresh pork versus nuts, beans, and eggs on postprandial plasma essential amino acid availability in older adults. Each participant will receive all four treatments.

DETAILED DESCRIPTION:
The 2015-2020 Dietary Guidelines for Americans (DGA) recommends how much protein-rich foods should be consumed as part of Healthy Eating Patterns. The predominant protein sources include lean meats, poultry, and eggs, along with nuts, seeds, and soy products (dairy is a separate category). Ounce-equivalent (oz-eq) is used as a standard unit of measure among these protein sources. One whole egg (1 oz-eq) is equal to 0.5 oz of nuts (1 oz-eq), 0.25 c (1 oz-eq) of beans, and 1 oz of lean meat (1 oz-eq). Importantly, protein quantity and quality of the foods are not considered. Consequently, consuming an oz-eq of protein foods from different sources may have different effects on an individuals' digestion, absorption, and use of the amino acids contained in proteins to build new proteins in their body (an anabolic response to feeding). Also importantly, while the current Recommended Dietary Allowance for protein (0.8 g total protein/kg/d) does not take into account the sources of protein consumed, these sources have varied essential amino acid patterns. The purpose of this study is to expand on a recent study assessing the effect of consuming ounce-equivalents of eggs versus pork, nuts, and beans on essential amino acid (EAA) substrate availability for protein anabolism in younger adults to include a cohort of older adults. Findings from this current research will allow direct comparisons of postprandial EAA substrate availability between different protein-rich food sources in a cohort of older adults (primary outcome). Subsequently, investigating postprandial responses of the same ounce-equivalents of fresh pork versus nuts, beans, and eggs on postprandial plasma essential amino acid availability in older adults will also allow for a comparison between the younger (from a study started prior to this one and still currently ongoing investigating the effect of the same ounce-equivalents of fresh pork versus nuts, beans, and eggs on postprandial plasma essential amino acid availability in adults) and older adult cohorts response to consuming different protein-rich foods (secondary outcome). This research will serve as an important resource for future DGA Committees to assess whether 'protein-ounce-equivalents' of varied protein-rich foods provide equivalent EAA substrate to promote postprandial protein synthesis in older adults, in support of dietary protein intake recommendations for younger and older adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 55-75
* BMI 20-35 kg∙m-2
* Weight stable (± 4.5 kg) 3 months pre-study
* Not acutely ill
* Not diabetic
* Not pregnant or lactating
* Not currently (or within 3 months pre-study) following a vigorous exercise regimen
* Non-smoking
* Willing to consume study foods and travel to testing facilities.

Exclusion Criteria:

-

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Plasma amino acid concentrations as measured by High Performance Liquid Chromatography (HPLC) | 5 hours
  Plasma samples will be drawn at times 0, 30, 60, 120, 180, 240, and 300 minutes after the consumption of the trial meal.
  The amino acids that will be assessed are alanine, arginine, asparagine, aspartic acid, cysteine, glutamic acid, glutamine, glycine, histidine, isoleucine, leucine, lysine, methionine, phenylalanine, proline, serine, threonine, tryptophan, tyrosine, valine.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States